CLINICAL TRIAL: NCT00654095
Title: Open-label, Long-term Study of Coadministration of Ezetimibe and Atorvastatin in Patients With Primary Hypercholesterolemia Who Have Not Reached LDL-cholesterol Target With HMG-CoA Reductase Inhibitors
Brief Title: Coadministration of Ezetimibe and Atorvastatin in Patients With Primary Hypercholesterolemia (P05456)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Organon and Co (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: P05456
Record Dates: First submitted 2008-04-01; First posted 2008-04-07 (Estimated); Results first posted 2010-10-05 (Estimated); Last update posted 2024-05-21 (Actual); Status verified 2022-02

CONDITIONS: Hypercholesterolemia
MeSH Terms: conditions — Hypercholesterolemia | interventions — Ezetimibe; Atorvastatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Ezetimibe + Atorvastatin (Experimental): Ezetimibe 10 mg + Atorvastatin 20 mg
  Interventions: Drug: Ezetimibe; Drug: atorvastatin

INTERVENTIONS:
Drug: Ezetimibe — Ezetimibe 10 mg once daily
  Other Names: SCH 58235
Drug: atorvastatin — atorvastatin 20 mg once daily

SUMMARY:
Evaluate the safety of the long-term (1 year) coadministration of ezetimibe and atorvastatin in participants with hypercholesterolemia who have not reached low density lipoprotein (LDL)-cholesterol target with 3-hydroxy-3-methylglutaryl-coenzyme A (HMG-CoA) reductase inhibitors.

ELIGIBILITY:
Inclusion Criteria:

* Participants with hypercholesterolemia who satisfy the following criteria:

  * Participants who have used any of the following 3-hydroxy-3-methylglutaryl-coenzyme A (HMG-CoA) reductase inhibitors (hereinafter referred to as "statins") for 4 weeks or longer before the start of the observation period and whose low density lipoprotein (LDL)-cholesterol level during the treatment had not reached lipid management target
  * Age: 20 years of age or older (at the time of obtaining informed consent)
  * Sex: both males and females
  * Inpatient/outpatient: Out-patient

Exclusion Criteria:

* Participants for whom any of the following is applicable:

  * Participants whose fasted triglyceride level measured at the start of the observation period or the treatment period exceeds 500 mg/dL
  * Participants with homozygous familial hypercholesterolemia
  * Participants with creatine phosphokinase (CPK) > 2x upper limit of normal (ULN) measured at the start of the observation period or the treatment period.
  * Participants with serious hepatic disorder, or participants with alanine aminotransferase (ALT) or aspartate aminotransferase (AST) > 2x ULN measured at the start of the observation period or the treatment period.
  * Participants with a history of hypersensitivity to any ingredient of ezetimibe tablets or atorvastatin tablets
  * Pregnant, nursing women, women who may be pregnant, or participants wishing to be pregnant during the study.
  * Participants who have discontinued use of serum lipid lowering agents for less than 4 weeks at the start of the treatment period (8 weeks in the case of probucol). (However, if the participant had taken a serum lipid lowering agent before the test conducted at the start of the observation period, a period of discontinuation of 27 days, or 55 days in the case of probucol, is allowed.)
  * Participants who are using cyclosporine from after the start of the observation period
  * Participants with a history of ezetimibe use
  * Participants with hyperlipidemia associated with the following diseases:

    * Hypothyroidism
    * Obstructive gall bladder or biliary disease
    * Chronic renal failure
    * Pancreatitis
  * Participants with hyperlipidemia associated with concomitant use of drugs having adverse effect on serum lipids, etc
  * Participants who have received an investigational drug within 4 weeks of the start of the observation period
  * Other participants deemed not appropriate for study entry by the investigator

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 146 (Actual)
Dates: Start 2007-12-01 (Actual); Primary Completion 2009-06-01 (Actual); Study Completion 2009-06-01 (Actual)

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Participants did not Complete the Study:
  1. level below what was specified in inclusion criterion
  2. level >500 mg/dL at start of treatment
  3. level >2x upper limit of normal at start of treatment
  4. level >=3x upper limit of normal after start of treatment
  5. Adverse reactions did not improve or resolve after dose reduction of atorvastatin
Groups:
- Ezetimibe + Atorvastatin: Ezetimibe 10 mg once daily + Atorvastatin 20 mg once daily
Period: Overall Study
Arm/Group | Ezetimibe + Atorvastatin
Started | 146
Completed | 114
Not Completed | 32
Not completed — Drop in low density lipoprotein (1) | 2
Not completed — Elevated triglyceride level (2) | 1
Not completed — Elevated alanine aminotransferase (3) | 1
Not completed — Adverse Event | 11
Not completed — Withdrawal by Subject | 5
Not completed — Elevated alanine aminotransferase (4) | 7
Not completed — Adverse reaction did not improve (5) | 4
Not completed — Did not meet inclusion criteria | 1

BASELINE CHARACTERISTICS:
Arm/Group | Ezetimibe + Atorvastatin
Number analyzed (Participants) | 146
Age, Customized [Number; unit: Participants] — >=20 Years
  Participants | 146
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 79
  Male | 67
Region of Enrollment [Number; unit: participants]
  Japan | 146

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Adverse Events and Adverse Reactions
Description: An adverse event is any unfavorable medical event occurring in a subject to whom an investigational product is administered, and a causal relationship between the administered investigational product and an adverse event is not always clarified.
  That is, an adverse event is any unfavorable or unintended sign (including an abnormal change in laboratory test values), symptom, or disease, and a causal relationship to the relevant investigational product is not considered.
  Any adverse event that was considered treatment-related was considered an adverse reaction.
Time Frame: Throughout 1 year of study
Measure: Number; unit: Participants
Arm/Group | Ezetimibe + Atorvastatin
Number analyzed (Participants) | 146
Participants
  Adverse Events | 141
  Adverse Reactions | 61

ADVERSE EVENTS:
Arm/Group | Ezetimibe+Atorvastatin
Serious Adverse Events (participants affected / at risk) | 11/146
Other Adverse Events (participants affected / at risk) | 132/146
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ezetimibe+Atorvastatin (N=146)
SICK SINUS SYNDROME (Cardiac disorders) | 1 (1)
GLAUCOMA (Eye disorders) | 1 (1)
RETINAL ARTERY OCCLUSION (Eye disorders) | 1 (1)
GASTROENTERITIS (Infections and infestations) | 1 (1)
HUMERUS FRACTURE (Injury, poisoning and procedural complications) | 1 (1)
IN-STENT CORONARY ARTERY RESTENOSIS (Injury, poisoning and procedural complications) | 1 (1)
RIB FRACTURE (Injury, poisoning and procedural complications) | 1 (1)
ULNA FRACTURE (Injury, poisoning and procedural complications) | 1 (1)
BREAST CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
LYMPHOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
PANCREATIC NEOPLASM (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
PROSTATE CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
CEREBRAL HAEMORRHAGE (Nervous system disorders) | 1 (1)
BENIGN PROSTATIC HYPERPLASIA (Reproductive system and breast disorders) | 1 (1)
ERYTHEMA MULTIFORME (Skin and subcutaneous tissue disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ezetimibe+Atorvastatin (N=146)
CONSTIPATION (Gastrointestinal disorders) | 10 (10)
GASTRITIS (Gastrointestinal disorders) | 10 (11)
MALAISE (General disorders) | 10 (16)
SEASONAL ALLERGY (Immune system disorders) | 8 (9)
BRONCHITIS (Infections and infestations) | 11 (11)
GASTROENTERITIS (Infections and infestations) | 9 (11)
NASOPHARYNGITIS (Infections and infestations) | 53 (97)
PHARYNGITIS (Infections and infestations) | 8 (12)
ALANINE AMINOTRANSFERASE INCREASED (Investigations) | 48 (59)
ASPARTATE AMINOTRANSFERASE INCREASED (Investigations) | 16 (18)
BILIRUBIN CONJUGATED INCREASED (Investigations) | 18 (26)
BLOOD BILIRUBIN INCREASED (Investigations) | 11 (16)
BLOOD CREATINE PHOSPHOKINASE INCREASED (Investigations) | 20 (24)
C-REACTIVE PROTEIN INCREASED (Investigations) | 31 (39)
GAMMA-GLUTAMYLTRANSFERASE INCREASED (Investigations) | 24 (26)
GLYCOSYLATED HAEMOGLOBIN INCREASED (Investigations) | 9 (9)
MYOGLOBIN BLOOD INCREASED (Investigations) | 17 (23)
MYOGLOBIN URINE PRESENT (Investigations) | 17 (18)
WEIGHT INCREASED (Investigations) | 9 (9)
WHITE BLOOD CELL COUNT INCREASED (Investigations) | 11 (13)
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 11 (11)
BACK PAIN (Musculoskeletal and connective tissue disorders) | 12 (15)
MUSCULOSKELETAL STIFFNESS (Musculoskeletal and connective tissue disorders) | 8 (8)
HEADACHE (Nervous system disorders) | 8 (9)
RHINITIS ALLERGIC (Respiratory, thoracic and mediastinal disorders) | 10 (12)
UPPER RESPIRATORY TRACT INFLAMMATION (Respiratory, thoracic and mediastinal disorders) | 18 (23)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Principal Investigator (PI) agrees, for a period of 5 years following the Effective Date, to retain the Disclosure made to it by or on behalf of Sponsor (SPKK), in confidence and not to disclose it to any third party.

PI further agrees that during such time period it will not, either directly or indirectly, use the Disclosure for any purpose(s) other than that indicated herein without the prior written consent of SPKK.